CLINICAL TRIAL: NCT01237288
Title: Therapeutic Use of Oral Sodium Phosphate (Z-521) in Primary Hypophosphatemic Rickets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10010301
Record Dates: First submitted 2010-11-07; First posted 2010-11-09 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Primary Hypophosphatemic Rickets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Z-521 (Experimental)
  Interventions: Drug: Z-521

INTERVENTIONS:
Drug: Z-521

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of oral phosphate (Z-521) in subjects with primary hypophosphatemic rickets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as primary hypophosphatemic rickets based on familial history, genetic test or laboratory test results.

Exclusion Criteria:

* A hyperparathyroidism

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Serum ALP level | 6 month
Serum phosphate level | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Keiichi Ozono, M.D., Ph.D., Study Chair — Osaka University Hospital
Locations (4):
- Japan (4):
  - Chiba Children's Hospital, Chiba
  - Kanagawa Children's Medical Center, Kanagawa
  - Osaka University Hospital, Osaka
  - Tokyo Metropolitan Children's Medical Center, Tokyo

REFERENCES:
- [Derived] Ozono K, Hasegawa Y, Minagawa M, Adachi M, Namba N, Kazukawa I, Kitaoka T, Asakura Y, Shimura A, Naito Y. Therapeutic use of oral sodium phosphate (phosribbon((R)) combination granules) in hereditary hypophosphatemic rickets. Clin Pediatr Endocrinol. 2014 Jan;23(1):9-15. doi: 10.1292/cpe.23.9. Epub 2014 Feb 3. PMID 24532956